CLINICAL TRIAL: NCT02486328
Title: The Effect of Different Sedation Regimes Administered by Anesthesiologists or Endoscopists on Cognitive Functions in Lower Gastrointestinal System Endoscopy
Brief Title: The Effect of Different Sedation Regimes on Cognitive Function in Lower Gastrointestinal System Endoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Perihan Ekmekçi, Associate Professor, Ufuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: UfukU
Record Dates: First submitted 2015-06-24; First posted 2015-07-01 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Gastrointestinal Dysfunction; Alteration of Cognitive Function
Keywords: Cognitive dysfunction; Colonoscopy; Sedation
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Midazolam; Meperidine; Remifentanil; Propofol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group MM (Other): 2 mg midazolam and 20mg meperidine given intravenously and additional 1-2mg midazolam and 20mg meperidine (wtih a maximum total of 5 mg midazolam and 50 mg meperidine) given when FPS greater than 3
  Interventions: Drug: Midazolam; Drug: Meperidine
- Group RP (Other): 100 mcg/kg/min propofol infusion and 1 mcg/kg remifentanil bolus administered and additional 0,5 mcg/kg remifentanil bolus given when FPS greater than 3
  Interventions: Drug: Remifentanil; Drug: Propofol

INTERVENTIONS:
Drug: Midazolam — Dosage adjustment
  Other Names: Versed
  Arms: Group MM
Drug: Meperidine — Dosage adjustment
  Other Names: Demerol
  Arms: Group MM
Drug: Remifentanil — Dosage adjustment
  Other Names: Ultiva
  Arms: Group RP
Drug: Propofol — Dosage adjustment
  Other Names: Diprivan
  Arms: Group RP

SUMMARY:
There are different sedation regimes for lower gastrointestinal system endoscopy which can be administered by anesthesiologists and non-anesthesiologists. This study aims to compare the effects of propofol/remifentanil combination and midazolam/meperidine combination on early cognitive function following lower gastrointestinal system endoscopies.

DETAILED DESCRIPTION:
Sedation for lower gastrointestinal system endoscopies can be administered by anesthesiologists or endoscopists and cognitive dysfunction after this procedure has not been fully investigated. The aim of this study was to investigate the effect of different sedation regimes applied by anesthesiologists or endoscopists on early cognitive dysfunction. Following ethics committee approval and written informed consent, 100 patients were randomly divided into two groups. In Group MM where drug regime was solely determined by endoscopists, 2 mg midazolam and 20mg meperidine was given intravenously and additional 1-2mg midazolam and 20mg meperidine (wtih a maximum total of 5 mg midazolam and 50 mg meperidine) was given when facial pain scale (FPS) was greater than 3. In Group RP where drug regime was solely determined by anesthesiologists, 100 mcg/kg/min propofol infusion and 1 mcg/kg remifentanil bolus was administered and additional 0,5 mcg/kg remifentanil bolus was given when FPS was greater than 3. Bispectral index (BIS) and hemodynamic monitorization was carried out throughout the procedure and BIS 60-80 with FPS<3 was targeted. The time to Observer Assessment of Alertness/Sedation Scale (OAAS) score to reach 3 was measured after the procedure and Trieger Dot Test (TDT) and Digit Symbol Substitution Test (DSST) was repeated at 5th, 15th and 30th minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-65 years of age (ASA I-III risk groups), scheduled for elective colonoscopy

Exclusion Criteria:

* Patient refusal
* Mini mental test (MMT) score<26
* Amsterdam Preoperative Anxiety and Information Scale (APAIS ) score >10
* Advanced cardiopulmonary or psychiatric disease
* Chronic alcohol abuse
* Morbid obesity
* Known allergy to study drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2015-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Perihan Ekmekçi, Assoc Prof, Principal Investigator — Ufuk University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cohen LB, Dubovsky AN, Aisenberg J, Miller KM. Propofol for endoscopic sedation: A protocol for safe and effective administration by the gastroenterologist. Gastrointest Endosc. 2003 Nov;58(5):725-32. doi: 10.1016/s0016-5107(03)02010-8. PMID 14595310
- [Result] Ferreira AO, Cravo M. Sedation in gastrointestinal endoscopy: Where are we at in 2014? World J Gastrointest Endosc. 2015 Feb 16;7(2):102-9. doi: 10.4253/wjge.v7.i2.102. PMID 25685266
- [Result] Padmanabhan U, Leslie K, Eer AS, Maruff P, Silbert BS. Early cognitive impairment after sedation for colonoscopy: the effect of adding midazolam and/or fentanyl to propofol. Anesth Analg. 2009 Nov;109(5):1448-55. doi: 10.1213/ane.0b013e3181a6ad31. Epub 2009 Jul 17. PMID 19617584

RESULTS

PARTICIPANT FLOW:
Groups:
- Group MM: 2 mg midazolam and 20mg meperidine given intravenously and additional 1-2mg midazolam and 20mg meperidine (wtih a maximum total of 5 mg midazolam and 50 mg meperidine) given when facial pain scale (FPS) greater than 3
  Midazolam: Dosage adjustment
  Meperidine: Dosage adjustment
Period: Overall Study
Arm/Group | Group MM | Group RP
Started | 52 | 51
Completed | 50 | 50
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group MM | Group RP | Total
Number analyzed (Participants) | 52 | 51 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 51 | 103
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (13.6) | 53.7 (10.4) | 55.6 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 14 | 35
  Male | 31 | 37 | 68
Race/Ethnicity, Customized [Number; unit: participants] | 52 | 51 | 103
Region of Enrollment [Number; unit: participants]
  Turkey | 52 | 51 | 103
Weight [Mean (Standard Deviation); unit: kilograms] | 71.7 (11.7) | 73.1 (15.5) | 72.4 (13.8)
Mini Mental Test [Mean (Standard Deviation); unit: units on a scale] — A test consisting of 11 questions, range is 0 (worst)-30 (best). A score of 23 and lower is considered as cognitive impairment
  units on a scale | 28.2 (1.3) | 28.6 (1.6) | 28.3 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognitive Function
Description: As measured by Trieger Dot Test. The test does not have an upper limit; the time taken to complete the test is added to the number of dots missed by the patient and a result is obtained. The lowest score possible is 0. Higher values represent worse outcomes.
Time Frame: Baseline and 5, 15, 30 minutes after the procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group MM | Group RP
Number analyzed (Participants) | 50 | 50
units on a scale
  5th minute | 47.5 (10.6) | 40.4 (6.8)
  15th minute | 44.7 (9.2) | 37.8 (5.6)
  30th minute | 42 (7.9) | 35.4 (6)
Statistical Analysis 1: Comparison: Group MM vs Group RP; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change in Cognitive Function
Description: As measured by Digit Symbol Substitution Test. Scale range 0-9. No cut-off value. Higher results represent better outcomes
Time Frame: Baseline and 5, 15, 30 minutes after the procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group MM | Group RP
Number analyzed (Participants) | 50 | 50
units on a scale
  5th minute | 1.6 (1.2) | 2 (1.6)
  15th minute | 2.1 (1.4) | 2.8 (1.8)
  30th minute | 2.4 (1.4) | 3.5 (2.1)
Statistical Analysis 1: Comparison: Group MM vs Group RP; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Visual Analogue Scale Scores From the Baseline
Description: Pain as measured by Visual Analogue Scale. Range 1-10. No cut-off value, Higher results represent worse outcomes
Time Frame: Baseline and 5, 15, 30 minutes after the procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group MM | Group RP
Number analyzed (Participants) | 50 | 50
units on a scale
  5 minutes after the procedure | 0.9 (2.1) | 0.4 (1.1)
  15 minutes after the procedure | 0.5 (1.2) | 0.4 (1.1)
  30 minutes after the procedure | 0.1 (0.3) | 0.1 (0.7)
Statistical Analysis 1: Comparison: Group MM vs Group RP; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Heart Rate
Description: Heart rate as measured in beats per minute
Time Frame: Baseline and 1,2,3,5,10,15 and 20 minutes
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Group MM | Group RP
Number analyzed (Participants) | 50 | 50
beats per minute
  baseline | 90.2 (15.5) | 82.6 (10)
  1 minute in procedure | 89.6 (17.8) | 81.3 (11.3)
  2 minute in procedure | 88 (16.4) | 76 (11.7)
  3 minute in procedure | 87.6 (14.8) | 69.9 (8.6)
  5 minute in procedure | 87.7 (14.8) | 70.3 (8.9)
  10 minute in procedure | 85.3 (16.1) | 70 (8.9)
  15 minute in procedure | 85.4 (15) | 71.6 (9.6)
  20 minute in procedure | 85 (14.1) | 73.1 (9.8)
Statistical Analysis 1: Comparison: Group MM vs Group RP; Test type: Superiority or Other; p = 0.001, Kruskal-Wallis

5. Secondary Outcome: Mean Arterial Pressure
Description: mean arterial blood pressure as measured in mmHg
Time Frame: Baseline and 1,2,3,5,10,15 and 20 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Group MM | Group RP
Number analyzed (Participants) | 50 | 50
mmHg
  baseline | 105.7 (19.5) | 113.1 (13)
  1 minute in procedure | 103 (16.7) | 104 (14.4)
  2 minute in procedure | 104.5 (16.2) | 92.9 (11.9)
  3 minute in procedure | 105.8 (17.7) | 89.3 (15.9)
  5 minute in procedure | 101.5 (20.4) | 87.1 (14.3)
  10 minute in procedure | 103.8 (16.6) | 100 (15)
  15 minute in procedure | 102.4 (17.2) | 91.6 (18.5)
  20 minute in procedure | 99.3 (18.7) | 94.3 (15.8)
Statistical Analysis 1: Comparison: Group MM vs Group RP; Test type: Superiority or Other; p = 0.001, Kruskal-Wallis

6. Secondary Outcome: Peripheral Oxygen Saturation
Description: peripheral oxygen saturation as measured by pulse oximeter. Units are percentages, Scale range 0-100.
Time Frame: Baseline and 1,2,3,5,10,15 and 20 minutes
Measure: Mean (Standard Deviation); unit: Percent of oxygenated hemoglobin
Arm/Group | Group MM | Group RP
Number analyzed (Participants) | 50 | 50
Percent of oxygenated hemoglobin
  baseline | 97.2 (1.9) | 98.6 (0.9)
  1 minute in procedure | 97.2 (2) | 98 (2.2)
  2 minute in procedure | 97.5 (1.7) | 98.5 (0.9)
  3 minute in procedure | 97.6 (1.3) | 98.4 (1.1)
  5 minute in procedure | 97.4 (1.6) | 97.1 (4)
  10 minute in procedure | 97.2 (2.4) | 98.1 (1.3)
  15 minute in procedure | 97.2 (1.6) | 98.3 (1.1)
  20 minute in procedure | 97.4 (1.8) | 98.2 (2.2)
Statistical Analysis 1: Comparison: Group MM vs Group RP; Test type: Superiority or Other; p = 0.001, Kruskal-Wallis

ADVERSE EVENTS:
Arm/Group | Group MM | Group RP
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No